CLINICAL TRIAL: NCT06298877
Title: Frailty, Quality Of Life and Early Reversal of Temporary Defunctioning Stoma in Ovarian Cancer (FOLERO) : A Prospective Cohort Study to Determine the Effect of Frailty on Survival and to Assess Early Reversal of Temporary Intestinal Stoma
Brief Title: Frailty, Quality Of Life and Early Reversal of Temporary Defunctioning Stoma in Ovarian Cancer
Acronym: FOLERO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahar Salehi (Other)
Responsible Party: Sponsor-Investigator, Sahar Salehi, MD, Associate Professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-04696-01
Record Dates: First submitted 2024-02-26; First posted 2024-03-07 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Frailty (Experimental): Single arm study evaluating frailty by assessment of questionnaires and three different frailty tools
  Interventions: Other: Frailty and Quality of Life evaluation

INTERVENTIONS:
Other: Frailty and Quality of Life evaluation — Frailty and Quality of Life evaluation after surgery

SUMMARY:
Complete macroscopic surgical resection (CMR) requires extensive surgery and combined with chemotherapy confers best chance of survival in advanced ovarian cancer. During cytoreductive surgery 11% of women require a temporary diverting intestinal stoma.

Unexpectedly, our results from a unique fully accounted for population demonstrate that survival was not improved when increasing the proportion of women in whom CMR was achieved and in a yet unidentified subgroup of women extensive surgery was detrimental. In these women surgical treatment should be omitted in favor of chemotherapy only. Accordingly, there is an imperative need to improve patient selection to surgical treatment.

In Sweden, we treat an unselected population of women in a public healthcare system, where 30% of women with are >75 years. Despite these circumstances guidelines on patient-selection are lacking.

Age is an imprecise variable to base clinical decisions on but must be considered with an aging population. The dynamics between physiological changes of aging, comorbidity and medical condition are included in the concept of frailty, that has gained little attention in oncology, despite their potential to stratify risk and mortality.

The FOLERO study is a prospective adequately powered national cohort study with aim to determine if frailty instruments may be used to select patient to surgical treatment. In addition, we test the feasibility of early stoma reversal after index cytoreductive surgery in a small phase I trial and follow our patients Health Related Quality of Life after state of the art surgical treatment.

DETAILED DESCRIPTION:
Hypothesis: Frailty is a predictor of poor survival Primary objective: To assess three different frailty instruments as predictors of survival Exposure: Frailty according to the three different frailty instruments evaluated Control: No frailty according to the three different frailty instruments evaluated Primary outcome measure: Overall survival

Secondary objectives (selection):

* To evaluate the effect of sarcopenia on postoperative outcome and survival
* To evaluate the effect of surgical extent on postoperative outcome and survival
* To describe the HRQoL and symptoms of the" Low anterior resection syndrome" after surgery

Phase I sub-study on the feasibility and safety of early stoma reversal (Karolinska University Hospital only)

Hypothesis: Early stoma reversal in select patients with advanced ovarian cancer is feasible and safe.

Primary objective: To assess the feasibility and safety of early closure of defunctioning stoma after upfront cytoreductive surgery in ovarian cancer Primary outcome measure : Feasibility and safety of early stoma reversal as measured by rate of anastomotic leakage, urgent re- operations and time-interval to adjuvant chemotherapy (defined cut-offs based on historic comparison in the study protocol)

ELIGIBILITY:
Inclusion Criteria:

* Women with epithelial ovarian cancer scheduled for cytoreductive surgery with curative intent
* Age ≥18 years
* Signed written informed consent

Exclusion Criteria:

* Not able to understand the Swedish or English language
* Other diagnosis than ovarian cancer on final pathology

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2029-03-28 (Estimated); Study Completion 2029-03-28 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 24 months after index surgery
  Overall survival time is calculated from the date of index surgery to the date of death (due to any cause), or for patients still alive to the date of last follow-up.

SECONDARY OUTCOMES:
1-year mortality | 12 months from index surgery
  Mortality within 1-year after index surgery
Health related quality of life (HRQoL) (QLQ-C30) | At baseline, 12-15 weeks after index surgery and 12 months after index surgery
  Assessed by validated questionnaire and comprise the European Organisation for Research and Treatment of Cancer (EORTC), Core Questionnaire (QLQ-C30)
Health related quality of life (HRQoL) (QLQ-OV28) | At baseline, 12-15 weeks after index surgery and 12 months after index surgery
  Assessed by validated questionnaire and comprise the European Organisation for Research and Treatment of Cancer (EORTC), EORTC Quality of life Questionnaire Ovarian Cancer Module (QLQ)-OV28
Health related quality of life (HRQoL) (QLQ-ELD14) | At baseline, 12-15 weeks after index surgery and 12 months after index surgery
  Assessed by validated questionnaire and comprise the European Organisation for Research and Treatment of Cancer (EORTC), EORTC Quality of life Questionnaire Elderly Module (EORTC-QLQ-ELD14)
Health related quality of life (HRQoL) (EQ-5D-5L) | At baseline, 12-15 weeks after index surgery and 12 months after index surgery
  Assessed by validated questionnaire and comprise the European Organisation for Research and Treatment of Cancer (EORTC), EQ-5D-5L
Low anterior resection syndrome (LARS) | At baseline, 12-15 weeks after index surgery and 12 months after index surgery
  Assessed by the validated LARS questionnaire
Postoperative complications | 30 days after index surgery
  Assessed by validated instruments, Clavien-Dindo Classification
Readmissions | 30 days after index surgery
  Assessed by review of hospital records from the day of discharge after index surgery
Length of hospital stay | From date of index surgery to the date of discharge or at latest 90 days after index surgery
  Assessed by review of hospital records
Extent of surgery vs survival | Up to 60 months after index surgery
  Measured by surgical complexity score (as defined by the Mayo and Karolinska Surgical Complexity scores) and Peritoneal Cancer Index (PCI) both by assessment at the preoperative multidisciplinary conference
  The agreement between preoperative and peroperative assessment of surgical extent needed to achive complete macroscopic resection.
Sarcopenia vs post-operative outcome | Up to 60 months after index surgery
  Sarcopenia is measured by computed tomography and different muscle groups by different software programs (e.g. Coreslicer, Slice-o-matic etc.).
Standard regimen of adjuvant chemotherapy | At 1 year after index surgery
  Standard regimen of adjuvant chemotherapy is defined as Carboplatin (AUC 5) and Paclitaxel (175 mg/m2) every 21 days for 6 cycles. Dose and frequency will be assessed by review of hospital records
Time interval to adjuvant chemotherapy | From index surgery to first infusion of adjuvant chemotherapy
  Assessed by review of hospital records.
Total number of hospital days and readmissions within90 days after index surgery | 90 days after index surgery
  Total number of hospital days within 90 days after index surgery by review of hospital records
Health economics | At baseline, 12-15 weeks after index surgery and 1 year after index surgery
  Health economics will be assessed by the Eq5D-5L validated instrument
Recurrence or progression free survival | Up to 60 months after index surgery
  Defined as the time interval between index surgery and the date of recurrence or death, whichever comes first. For event-free patients recurrence free survival is the time between index surgery and the date for the last follow-up visit by review of medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Salehi, MD, PhD, Study Director — Karolinska University Hospital
Locations (4):
- Sweden (4):
  - Karolinska University Hospital, Stockholm, Solna
  - Sahlgrenska University Hospital and Sahlgrenska Academy, Gothenburg
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Lund

REFERENCES:
- [Derived] Hunde D, Ekerstad N, Asp M, Kannisto P, Wedin M, Palmqvist C, Dahm-Kahler P, Brandberg Y, Abraham-Nordling M, Ahlund K, Morlin V, Groes-Kofoed N, Salehi S. Determining the effect of frailty on survival in advanced ovarian cancer: study protocol for a prospective multicentre national cohort study (FOLERO). Acta Oncol. 2025 Feb 5;64:208-213. doi: 10.2340/1651-226X.2025.42292. PMID 39907536